CLINICAL TRIAL: NCT07327528
Title: Monocentric Pilot Study for the Application of an Endourethral Device for the Treatment of Stress Urinary Incontinence
Acronym: CIP-003
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Relief srl (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIP-003
Record Dates: First submitted 2025-08-05; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Urinary Incontinence , Stress
Keywords: Urinary incontinence, Stress
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic surgery for device installation (Experimental): Endoscopic surgery for device installation
  Interventions: Device: UroRelief, a sterile, single-use, endourethral medical device suitable for both men and women, which is positioned at the bladder neck for the treatment of stress incontinence.

INTERVENTIONS:
Device: UroRelief, a sterile, single-use, endourethral medical device suitable for both men and women, which is positioned at the bladder neck for the treatment of stress incontinence. — UroRelief is a sterile, single-use, endourethral medical device suitable for both men and women, which is positioned at the bladder neck for the treatment of stress incontinence. The device is designed to be inserted through the urethra using a routine endoscopic procedure with a resectoscope. Once in place, the device is completely inside the body with no visible parts outside and can restore urinary continence control.

SUMMARY:
Stress urinary incontinence is defined as the involuntary loss of urine during exertion or physical activity (i.e., sports) or during sneezing or coughing. Approximately 127 million women and 10 million men reported suffering from stress urinary incontinence in 2008, and current estimates are on the rise.

The prevalence of stress urinary incontinence is higher in older age groups, with 10% of women and 5% of men over the age of 65 suffering from this condition. The initial management of urinary incontinence consists of basic diagnostic investigations to rule out any reversible conditions (i.e., bacterial urinary tract infections, UTIs), while conservative and non-invasive treatment options include lifestyle changes, (PFMT) with or without biofeedback, and bladder retraining.

DETAILED DESCRIPTION:
Stress urinary incontinence is defined as the involuntary loss of urine during exertion or physical activity (i.e., sports) or during sneezing or coughing.

It is estimated to be the most common type of urinary incontinence worldwide due to its high prevalence in women. Approximately 127 million women and 10 million men reported suffering from stress urinary incontinence in 2008, and current estimates are on the rise. It can be primary or secondary and is caused by damage to either the sphincter innervation or the anatomical structures that make up the urethral sphincter. It is usually classified according to its severity and, consequently, according to the impairment of the patient's quality of life. It can seriously affect patients' quality of life in severalareas, leading to conditions such as sexual dysfunction, social isolation, withdrawal from physical activity, and major depression. The initial management of urinary incontinence consists of basic diagnostic investigations to rule out any reversible conditions (i.e., bacterial urinary tract infections, UTIs), while conservative and non-invasive treatment options include lifestyle changes, pelvic floor muscle training (PFMT) with or without biofeedback and bladder retraining, as well as the chronic and daily use of external aids (diapers).

The goal of treatment is to achieve complete or partial continence, with the aim of restoring normal sexual function. (PFMT) with or without biofeedback and bladder retraining, as well as the chronic and daily use of external aids (diapers, collection systems, prophylactics, etc.). However, this does not guarantee the restoration of a good quality of life. The current guidelines of the European Association of Urology (EAU) recommend surgical treatment when conservative and pharmacological therapies fail. In men, the most common surgical treatment for stress urinary incontinence that does not respond to therapy is the implantation of an artificial urethral sphincter, while in women, the indication is for complicated stress urinary incontinence (failure of other treatments such as retropubic or transobturator mid-retral slings). Currently, the most widely used device is a three-chamber device (consisting of a cuff, a balloon, and a pump) placed extraurethrally, whose application requires general and/or spinal anesthesia. The system proposed in the study, on the other hand, is an endourethral device to be applied endoscopically after anesthesia. The device is applied through a simple endoscopic maneuver without the need for other devices implanted in other anatomical sites and can be activated by slight abdominal pressure exerted by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (both women and men) aged between 21 and 85 years
* Documented stress urinary incontinence (urethral hypermobility or intrinsic sphincter deficiency) in which urgency symptoms are a minor component of the incontinence symptoms
* Stress urinary incontinence present and physiologically stable over the last 6 months.
* Urinary leakage >150 ml in the 24-hour PAD test performed during the pre-implantation screening phasefor male patients.- Urinary leakage >150 ml in the 24-hour PAD test performed during the pre-implantation screening phase
* Cognitive/manual ability to use the device.
* The patient is willing and able to meet the requirements of the protocol.
* The patient has decided to be implanted with the device for the treatment of urinary incontinence
* Willingness to sign the informed consent form.
* Willingness to return for follow-up evaluations and complete questionnaires.
* The patient has been informed about alternative therapies available for the treatment or management of urinary incontinence and about all possible risks associated with the implantation of the device.
* Any pre-existing urological conditions have been treated and resolved or are under control.
* Urinalysis and urine culture negative for infections and (micro)hematuria.
* Flexible cystoscopy with evidence of sphincter incompetence.

Exclusion Criteria:

* Primary urge incontinence or mixed stress and urge incontinence in which urge symptoms are a major component of the incontinence symptoms.
* Detrusor overactivity.
* History of recurrent bladder stones.
* Atonic neurogenic bladder or detrusor sphincter dyssynergia.
* Patients taking specific medications for bladder dysfunction or currently undergoing treatment for incontinence.
* Post-void residual urine >200 ml.
* Maximum cystometric capacity <150 ml.
* Detrusor pressure >20 cmH2O.
* Flexible cystoscopy showing stenosis that prevents device implantation.
* History of previously undiagnosed and unidentified microhematuria.
* Unexplained cystoscopic abnormalities and any suspected ongoing urological pathology.
* Asymptomatic bacteriuria during the screening period.
* History of bladder or upper urinary tract infections more than twice in the last 12 months.
* Patients requiring frequent catheterization or intermittent cystoscopy due to previous conditions.
* Female patients who are pregnant or planning to become pregnant within the next year.
* Stage II uterine prolapse in female patients.
* Previous pelvic surgery or radiotherapy in female patients.
* Any previous implantation of medical devices for urinary incontinence.
* History of sensitivity to silicone, titanium, nickel, and all materials listed in the technical data sheet.
* Vulnerable patients or those in emergency circumstances.
* The patient's health status precludes completion of follow-up, including terminal illnesses.
* Not willing/able to comply with the study requirements.
* Participation in any clinical study in the last 3 months.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-07-09 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The safety of UroRelief | 18 months
  - Complete characterization of all serious and unrecorded adverse events, including frequency and severity, reported throughout the study, according to the Clavien Dindo classification (I, II, 111°, IIIb, IVa, IVb, V).
The safety of UroRelief | 18 months
  - Pain assessed using the Visual Analog Scale (VAS) 1-10 for pain [Observation period:Baseline, 10, 30, 60, 90, and 120 days].
The safety of UroRelief | 18 months
  - Quality of sexual life assessed using the Female Sexual Function Index (FSFI) for women [Observation period: Baseline, 10, 30, 60, 90, and 120 days].
The safety of UroRelief | 18 months
  - Quality of sexual life assessed using the International Index of Erectile Function (IIEF) questionnaire for men [Observation period: Baseline, 10, 30, 60, 90, and 120 days].

SECONDARY OUTCOMES:
Assess incontinence at 30 days, measured using the 24-hour pad weight test. | 18 months
  Percentage of patients with a significant reduction in incontinence at 60 days. A subject is considered a success if they experience a reduction in the weight of the diaper over 24 hours of at least 50% at 30 days compared to the baseline value.

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Grande Ospedale Metropolitano Niguarda, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided